CLINICAL TRIAL: NCT06083870
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Oba01 for Injection in Patients With DR5 Positive LA/mNSCLC
Brief Title: An Early Stage Study to Evaluate Oba01 for Injection in Patients With DR5 Positive LA/mNSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lu Shun (Other)
Responsible Party: Sponsor-Investigator, Lu Shun, Prof., Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC248-C001
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oba01 (Experimental)
  Interventions: Drug: Oba01

INTERVENTIONS:
Drug: Oba01 — Oba01 0.15, 0.5, 0.75, 1.0 mg/kg by intravenous (IV) infusion, given on Day 1 of each 21-day cycle

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and efficacy of Oba01 for injection in patients with DR5 positive LA/mNSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Man or woman ≥ 18 years and ≤75 years of age at the time of enrollment.
* Histologically and/or cytologically-confirmed locally advanced or metastatic NSCLC.
* Measurable lesion according to RECIST 1.1.
* Progression after systemic treatment for advanced NSCLC.
* Available archived paraffin-embedded or fresh tumor tissue from the primary tumor or metastasis for submission to the central laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Measurable and/or non-measurable disease as per RECIST 1.1 criteria.
* Adequate organ function as assessed by laboratory tests.
* Male or female subjects of child-producing potential must agree to use avoidance of pregnancy measures during the study and for 6 months after the last day of treatment.

Exclusion Criteria:

* Patient has received previous treatment with DR5 targeted regimen or antibody-MMAE conjugate.
* Brain metastases unless asymptomatic, stable and not requiring steroids for at least 7 days prior to start of study treatment.
* Subject with positive HCV-Ab, Anti-HIV or positive HBS-Ag with copies of HBV DNA > ULN.
* Pregnancy, lactation, or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
maximal tolerance dose (MTD) of Oba01 | DLT will be evaluated on 21 days of observation period
  Maximum-tolerated dose (MTD) was defined as the highest dose level at which no more than one of six patients experienced DLT during the DLT assessment window.

SECONDARY OUTCOMES:
Overall response rate(ORR) | Up to approximately 2 years
  The objective response rate will be mainly analyzed by investigators according to the RECIST 1.1 standard tumor evaluation.
Disease control rate (DCR) | Up to approximately 2 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study.
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) refers to the time from the date of first dose to the first researcher's evaluation of disease progression or death.
Overall survival (OS) | Up to approximately 2 years
  Overall survival (OS) refers to the time from the date of first dose to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Shanghai Lung Cancer Center, Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No